CLINICAL TRIAL: NCT00618033
Title: Short-Term Study of Physiologic Dialysate Glucose Concentration in Chronic Hemodialysis Patients
Brief Title: Comparison of Different Glucose Concentrations in Dialysate of Hemodialysis Patients
Acronym: Dextrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renal Research Institute (Other)
Responsible Party: Nathan Levin, MD, Renal Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 169-07
Record Dates: First submitted 2008-02-04; First posted 2008-02-18 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Hemodialysis; ESRD
Keywords: Hemodialysis; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Hemodialysis
- 2 (Active Comparator)
  Interventions: Procedure: Hemodialysis

INTERVENTIONS:
Procedure: Hemodialysis — varying concentration of glucose in dialysate

SUMMARY:
This study aims to show that using a glucose (sugar) concentration of 100 mg/dL in the dialysis fluid for hemodialysis is not inferior to using a concentration of 200 mg/dL with regard to the frequency and magnitude of blood glucose drops. Other parameters that will be compared between the two groups are blood pressure, heart rhythm, weight gain between dialysis treatments, and fatigue after the treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blinded cross-over non-inferiority trial of intra- and early post-dialytic glucose homeostasis comparing 100 mg/dL against 200 mg/dL dialysate glucose concentration in 30 hemodialysis patients. The primary outcome is the frequency and magnitude of hypoglycemia during and early after the hemodialysis treatment. Secondary outcomes include intradialytic blood pressure, interdialytic weight gain, serum potassium and phosphorus concentrations, arrhythmias during dialysis and in the early postdialytic period, and postdialytic fatigue.

Inclusion criteria:

Age ≥ 18 years

Maintenance hemodialysis with hemodialysis vintage of at least 30 days

Ability to read and understand the English language and give informed consent

Exclusion criteria:

Dialysis treatment frequencies other than three times per week

Hospitalizations or antibiotics-dependent infection during the 8 weeks preceding enrollment

Central venous catheter as hemodialysis access

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Maintenance hemodialysis with hemodialysis vintage of at least 30 days
* Ability to read and understand the English language and give informed consent

Exclusion Criteria:

* Dialysis treatment frequencies other than three times per week
* Hospitalisations or antibiotics-dependent infection during the 8 weeks preceding enrollment
* Central venous catheter as hemodialysis access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Frequency and magnitude of hypoglycemia during and early after the hemodialysis treatment | 6 weeks

SECONDARY OUTCOMES:
Intradialytic blood pressure, interdialytic weight gain, serum potassium and phosphorus concentrations, arrhythmias during dialysis and in the early postdialytic period, postdialytic fatigue | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathan W. Levin, MD, Principal Investigator — Renal Research Institute
Locations (2):
- United States (2):
  - Irving Place Dialysis Center, New York, New York
  - Yorkville Dialysis Center, New York, New York

REFERENCES:
- [Result] Raimann JG, Kruse A, Thijssen S, Kuntsevich V, Diaz-Buxo JA, Levin NW, Kotanko P. Fatigue in hemodialysis patients with and without diabetes: results from a randomized controlled trial of two glucose-containing dialysates. Diabetes Care. 2010 Sep;33(9):e121. doi: 10.2337/dc10-1043. No abstract available. PMID 20805263
- [Result] Ferrario M, Raimann JG, Thijssen S, Signorini MG, Kruse A, Diaz-Buxo JA, Cerutti S, Levin NW, Kotanko P. Effects of dialysate glucose concentration on heart rate variability in chronic hemodialysis patients: results of a prospective randomized trial. Kidney Blood Press Res. 2011;34(5):334-43. doi: 10.1159/000327851. Epub 2011 May 25. PMID 21613795
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Raimann JG, Kruse A, Thijssen S, Kuntsevich V, Dabel P, Bachar M, Diaz-Buxo JA, Levin NW, Kotanko P. Metabolic effects of dialyzate glucose in chronic hemodialysis: results from a prospective, randomized crossover trial. Nephrol Dial Transplant. 2012 Apr;27(4):1559-68. doi: 10.1093/ndt/gfr520. Epub 2011 Sep 22. PMID 21940484